CLINICAL TRIAL: NCT04628065
Title: #BabyLetsMove: A Feasibility Study of a mHealth Physical Activity Intervention for Perinatal Adolescents
Brief Title: #BabyLetsMove Physical Activity Feasibility Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Mississippi Medical Center (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH); Mississippi State Department of Health (Other Government)
Responsible Party: Principal Investigator, Abigail Gamble, Assistant Professor, University of Mississippi Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2017-0024; 1U54GM115428 (NIH)
Record Dates: First submitted 2020-10-30; First posted 2020-11-13 (Actual); Last update posted 2022-08-08 (Actual); Status verified 2022-08

CONDITIONS: Pregnancy Related; Adolescent Obesity; Behavior, Health; Behavior, Sedentary; Adolescent Overweight; Mobile Phone Use; Pregnancy in Adolescence
Keywords: Pregnancy in adolescence; Exercise; Physical activity; Sedentary behavior; mHealth; Obesity in pregnancy; Adolescent obesity; Adolescent overweight; Behavioral science; Implementation science; Clinical trial
MeSH Terms: conditions — Pediatric Obesity; Health Behavior; Sedentary Behavior; Cell Phone Use; Motor Activity; Pregnancy in Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention Arm (Experimental): Participants will receive a text message everyday to build behavioral skills and practice self-monitoring of three behavior goals: (1) reduce TV time to less than 2 hours per day; (2) take 10,000 steps or more every day; (3) do 20 minutes or more of structures exercise like prenatal yoga or dance videos every day. Participants will also receive two health coaching mobile phone session; an introduction session and one problem solving session.
  Interventions: Behavioral: #BabyLetsMove

INTERVENTIONS:
Behavioral: #BabyLetsMove — This intervention will use mobile phones to promote the adoption and maintenance of physical activity, exercise and reduced TV time among overweight or obese, Black, pregnant (<16 weeks) adolescents (15 - 19 years) enrolled in Mississippi's WIC program.

SUMMARY:
Black adolescents who are pregnant represent a high-risk and understudied perinatal population in health research. Adolescent pregnancy (<20 years) is disproportionately prevalent among Blacks compared with Whites and is a prominent risk factor for obesity. Fortunately, metabolic consequences of increasing physical activity coupled with minimal sedentary time can mitigate biological imperils and behavioral interventions targeting perinatal populations have demonstrated efficacy for this approach. Intervention studies to promote physical activity and reduce sedentarism among Black, perinatal adolescents in disadvantaged, rural settings may be a promising strategy to prevent obesity and reduce disparities. In the proposed study, investigators will assess the feasibility and acceptability of #BabyLetsMove, a mobile health intervention targeting three behavioral goals: (1) limit TV time to less than 2 hours a day (sedentary behavior); (2) take 10,000 steps or more per day (physical activity); and (3) do 20 minutes or more of structured activity like prenatal yoga or dance videos per day (exercise). In the #BabyLetsMove feasibility trial investigators aim to conduct a single-arm, 4-week pilot with 20 Black adolescents (15- to 19-years) enrolled in Mississippi's Supplemental Nutritional Program for Women, Infants and Children (WIC) to test the intervention's feasibility and acceptability. Participants will receive one text message per day for 4-weeks targeting behavior change strategies and two health coaching sessions via mobile phone; an introduction session in week one and a problem-solving session in week three. Investigators will also use qualitative interviewing with additional adolescents (n=20) to solicit user feedback regarding the acceptability of intervention content and materials. Finally, in preparation for a pilot study using an effectiveness-implementation hybrid study design, investigators will conduct a pre-implementation evaluation using quantitative surveying (n=6 surveys) with WIC providers (n=60) to better under the culture and climate of WIC. Investigators hypothesize the #BabyLetsMove intervention will be acceptable to adolescents and a future pilot randomized controlled trial will be feasible. Investigators also anticipate identifying modifiable barriers and facilitators to implementing the intervention through WIC, which will help to design an implementation strategy with a high likelihood for uptake by WIC.

DETAILED DESCRIPTION:
Formative research is needed to establish a foundation for obesity prevention research with high-risk, disadvantaged, perinatal adolescents and their offspring. In particular, Black pregnant adolescents in socioeconomically disadvantaged communities represent a high-risk and understudied perinatal population in health research. Adolescent pregnancy (<20 years) is disproportionately prevalent among Blacks compared with Whites (27.6 and 13.4 per 1,000, respectively) and is a prominent risk factor for obesity. Normal pubertal growth is associated with increased weight in adolescence and Black female and rural adolescents are at highest risk for excessive adiposity. Pregnancy exacerbates preexisting risks and predicates a trajectory of maternal and child obesity. Fortunately, metabolic consequences of increasing physical activity coupled with minimal sedentary behavior can mitigate biological imperils and behavioral interventions targeting perinatal populations have demonstrated efficacy for this approach. Intervention studies to promote physical activity and reduce sedentary behavior among Black, perinatal adolescents in disadvantaged, rural settings may be a promising strategy to prevent obesity and reduce disparities. To this end, investigators conducted formative work in the Teen Mom Study, an exploratory investigation to identify modifiable psychosocial, cultural and environmental determinants of physical activity among pregnant and postpartum adolescents enrolled in Mississippi's Supplemental Nutritional Program for Women Infants and Children (WIC) in the Mississippi Delta. WIC is a federally-funded, state-run public health service providing healthy food and nutrition counseling to low-income women, infants and children at nutritional risk. Public health services like WIC are ideal settings for the prevention and treatment of obesity among high-risk, socioeconomically disadvantaged populations. The Mississippi Delta is a culturally and geographically distinct 18-county rural region of Mississippi that is plagued by decades of persistent poverty, poor health and the highest teen birth rate, which has not declined since 2006, in the United States. Using data from the Teen Mom Study, investigators adapted an existing mobile health (mHealth) intervention to achieve three behavioral goals: (1) limit TV time to less than 2 hours a day (sedentary behavior); (2) take 10,000 steps or more per day (physical activity; tracked using a FitBit provided to each study participant); and (3) do 20 minutes or more of structured activity like prenatal yoga or dance videos per day (exercise). In the #BabyLetsMove feasibility trial investigators aim to conduct a single-arm, 4-week pilot with 20 overweight or obese, Black, pregnant (<16 weeks) adolescent (15 - 19 years) WIC clients to test the feasibility and acceptability of the intervention. Participants will receive text messages aligned with theoretical behavior change strategies every day of the week for 4-weeks including: 1) four skills texts, which may be a simple text or a text with a link to either a PDF or video; 2) two goal monitoring text messages, which will check-in on the three behavior change goals; and 3) and one text message for participants to report their weight using a BodyTrace scale provided by the study. Text messages will be supplemented with two health coaching telephone calls conducted by the principal investigator; an introduction session in the first week, followed by a problem-solving session in week three. While the study goal is to assess feasibility and acceptability, physical activity assessed using accelerometry, subjective psychosocial constructs, and anthropometric and biomarker measures will be measured at pre- (week 1) and post- (week 6) intervention. To gain additional insight, investigators will use qualitative interviewing with additional adolescents (n=20) to solicit user feedback regarding the acceptability of intervention content (text messages) and materials (PDFs and videos). Finally, in preparation for a randomized pilot trial using an effectiveness-implementation hybrid research design, investigators will conduct a pre-implementation evaluation using quantitative surveying (n=6 surveys) with WIC providers (n=60) to better under the context, culture and climate of WIC (implementation measures identified in the Consolidated Framework for Implementation Research). Investigators hypothesize the #BabyLetsMove intervention materials will be acceptable to adolescents and that conducting a future pilot randomized controlled trial will be feasible. Investigators also anticipate identifying modifiable barriers and facilitators to implementing the intervention through WIC, which will help to design an implementation strategy with a high likelihood for uptake by WIC. If proven to be effective, #BabyLetsMove mHealth intervention may be a scalable approach to increase physical activity among socioeconomically disadvantaged adolescents at high risk for maternal and child obesity.

ELIGIBILITY:
Inclusion Criteria:

* African American or Black
* <16 weeks gestation
* Overweight or obese
* Enrolled in WIC
* Resides in one of 13 Mississippi Delta Counties
* Cohabitation with their mother
* Has a personal smart phone

Exclusion Criteria:

* Been told by a doctor they can not exercise

Ages: 15 Years to 19 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 14 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Physical activity | Baseline, pre-intervention
  Objective physical activity assessed using Actigraph GT9X accelerometry worn for seven consecutive days
Sedentary time | Baseline, pre-intervention
  Objective physical activity assessed using Actigraph GT9X accelerometry worn for seven consecutive days

SECONDARY OUTCOMES:
Body weight | Baseline, pre-intervention
  BodyTrace scale with Bluetooth
Readiness for physical activity in pregnancy | Baseline, pre-intervention
  Single response item to categorize readiness to engage in physical activity; Haakstad et al., 2013 (PMID:23431448)
Self-efficacy for physical activity | Baseline, pre-intervention
  5-item survey to assess confidence in doing 20-minutes or more of moderate intensity on 1 day per week, 2 days, 3 days, 4 days, and 5 or more days; 11-point Likert scale from 0, absolutely not confident, to 100, absolutely confident
Self-efficacy for overcoming self-identified barriers to physical activity | Baseline, pre-intervention
  Up to 4-item instrument to list perceived barriers to physical activity and rating confidence to overcome each barrier using an 11-point Likert scale from 0, absolutely not confident, to 100, absolutely confident
Self-efficacy for limiting sedentary time | Baseline, pre-intervention
  6-item instrument to rate confidence in limiting sedentary time using an 11-point Likert scale from 0, absolutely not confident, to 100, absolutely confident;
Self-regulation: Goal-Setting | Baseline, pre-intervention
  Exercise Goal-Setting Scale; 10 items rated using a 5-point Likert scale from 1, does not describe me, to 5, describes me completely
Self-regulation: Planning | Baseline, pre-intervention
  Exercise Planning Scale; 10 items rated using a 5-point Likert scale from 1, does not describe me, to 5, describes me completely
Decisional balance | Baseline, pre-intervention
  Pros and Cons of Reducing TV Time; 11-items rated using 4-point Likert scale from 1, strongly disagree to 4, strongly agree
Perceived exercise safety in pregnancy | Baseline, pre-intervention
  Exercise Safety Scale; 14 items rated using a 4-point Likert scale from 1, very unsafe to 4, very safe
Perceived daily physical activity behavior | Baseline, pre-intervention
  Pregnancy Physical Activity Questionnaire; 32-item survey to assess type and duration of physical activities on a typical day within respective trimester using 6-point Likert scale from 0, non to 6, 3 or more hours per day

OTHER OUTCOMES:
Organizational Identification | Baseline, pre-intervention
  Organizational Identification Scale; 25-items rated using a 6-point Likert scale from 1, strongly disagree to 6, strongly agree
Inner Setting | Baseline, pre-intervention
  Inner Setting Measures from the Consolidated Framework for Implementation Research; 34-items rated using a 6-point Likert scale from 1, strongly disagree to 6, strongly agree
Organizational Climate | Baseline, pre-intervention
  Organizational Climate Survey; 28-items using a 6-point Likert scale from strongly disagree to 6, strongly agree
Psychosocial factors at work: quantitative demands | Baseline, pre-intervention
  Copenhagen Psychosocial Questionnaire (COPSOQ-II) long form; a battery of scales used in research to measure psychosocial factors at work (128-items total); 4-items using a 5-point Likert scale from 0, never to 100, always
Psychosocial factors at work: work pace | Baseline, pre-intervention
  Copenhagen Psychosocial Questionnaire (COPSOQ-II) long form; a battery of scales used in research to measure psychosocial factors at work (128-items total); 3-items using a 5-point Likert scale from 0, to a very small extent to 100, to a very large extent
Psychosocial factors at work: cognitive demands | Baseline, pre-intervention
  Copenhagen Psychosocial Questionnaire (COPSOQ-II) long form; a battery of scales used in research to measure psychosocial factors at work (128-items total); 4-items using a 5-point Likert scale from 0, never to 100, always
Psychosocial factors at work: emotional demands | Baseline, pre-intervention
  Copenhagen Psychosocial Questionnaire (COPSOQ-II) long form; a battery of scales used in research to measure psychosocial factors at work (128-items total); 4-items using a 5-point Likert scale from 0, never to 100, always
Psychosocial factors at work: demands for hiding emotions | Baseline, pre-intervention
  Copenhagen Psychosocial Questionnaire (COPSOQ-II) long form; a battery of scales used in research to measure psychosocial factors at work (128-items total); 3-items using a 5-point Likert scale from 0, never to 100, always
Psychosocial factors at work: influence | Baseline, pre-intervention
  Copenhagen Psychosocial Questionnaire (COPSOQ-II) long form; a battery of scales used in research to measure psychosocial factors at work (128-items total); 4-items using a 5-point Likert scale from 0, never to 100, always
Psychosocial factors at work: possibilities for development | Baseline, pre-intervention
  Copenhagen Psychosocial Questionnaire (COPSOQ-II) long form; a battery of scales used in research to measure psychosocial factors at work (128-items total); 4-items using a 5-point Likert scale from 0, to a very small extent to 100, to a very large extent
Psychosocial factors at work: variation of work | Baseline, pre-intervention
  Copenhagen Psychosocial Questionnaire (COPSOQ-II) long form; a battery of scales used in research to measure psychosocial factors at work (128-items total); 2-items using a 5-point Likert scale from 0, never to 100, always
Psychosocial factors at work: meaning of work | Baseline, pre-intervention
  Copenhagen Psychosocial Questionnaire (COPSOQ-II) long form; a battery of scales used in research to measure psychosocial factors at work (128-items total); 3-items using a 5-point Likert scale from 0, to a very small extent to 100, to a very large extent
Psychosocial factors at work: commitment to the workplace | Baseline, pre-intervention
  Copenhagen Psychosocial Questionnaire (COPSOQ-II) long form; a battery of scales used in research to measure psychosocial factors at work (128-items total); 4-items using a 5-point Likert scale from 0, to a very small extent to 100, to a very large extent
Psychosocial factors at work: predictability | Baseline, pre-intervention
  Copenhagen Psychosocial Questionnaire (COPSOQ-II) long form; a battery of scales used in research to measure psychosocial factors at work (128-items total); 2-items using a 5-point Likert scale from 0, to a very small extent to 100, to a very large extent
Psychosocial factors at work: rewards (recognition) | Baseline, pre-intervention
  Copenhagen Psychosocial Questionnaire (COPSOQ-II) long form; a battery of scales used in research to measure psychosocial factors at work (128-items total); 3-items using a 5-point Likert scale from 0, to a very small extent to 100, to a very large extent
Psychosocial factors at work: role clarity | Baseline, pre-intervention
  Copenhagen Psychosocial Questionnaire (COPSOQ-II) long form; a battery of scales used in research to measure psychosocial factors at work (128-items total); 3-items using a 5-point Likert scale from 0, to a very small extent to 100, to a very large extent
Psychosocial factors at work: role conflicts | Baseline, pre-intervention
  Copenhagen Psychosocial Questionnaire (COPSOQ-II) long form; a battery of scales used in research to measure psychosocial factors at work (128-items total); 4-items using a 5-point Likert scale from 0, to a very small extent to 100, to a very large extent
Psychosocial factors at work: perceived quality of leadership | Baseline, pre-intervention
  Copenhagen Psychosocial Questionnaire (COPSOQ-II) long form; a battery of scales used in research to measure psychosocial factors at work (128-items total); 4-items using a 5-point Likert scale from 0, to a very small extent to 100, to a very large extent
Psychosocial factors at work: social support from supervisor | Baseline, pre-intervention
  Copenhagen Psychosocial Questionnaire (COPSOQ-II) long form; a battery of scales used in research to measure psychosocial factors at work (128-items total); 3-items using a 5-point Likert scale from 0, never to 100, always
Psychosocial factors at work: social support from colleagues | Baseline, pre-intervention
  Copenhagen Psychosocial Questionnaire (COPSOQ-II) long form; a battery of scales used in research to measure psychosocial factors at work (128-items total); 3-items using a 5-point Likert scale from 0, never to 100, always
Psychosocial factors at work: social community at work | Baseline, pre-intervention
  Copenhagen Psychosocial Questionnaire (COPSOQ-II) long form; a battery of scales used in research to measure psychosocial factors at work (128-items total); 3-items using a 5-point Likert scale from 0, never to 100, always
Psychosocial factors at work: job insecurity | Baseline, pre-intervention
  Copenhagen Psychosocial Questionnaire (COPSOQ-II) long form; a battery of scales used in research to measure psychosocial factors at work (128-items total); 4-items using a 5-point Likert scale from 0, to a very small extent to 100, to a very large extent
Psychosocial factors at work: perceived job satisfaction | Baseline, pre-intervention
  Copenhagen Psychosocial Questionnaire (COPSOQ-11) long form; a battery of scales used in research to measure psychosocial factors at work (128-items total); 4-items using a 5-point Likert scale from 0, not relevant to 100, very satisfied
Psychosocial factors at work: work-family conflict | Baseline, pre-intervention
  Copenhagen Psychosocial Questionnaire (COPSOQ-II) long form; a battery of scales used in research to measure psychosocial factors at work (128-items total); 4-items using a 4-point Likert scale from 0, no not at all to 100, yes certainly
Psychosocial factors at work: family-work conflict | Baseline, pre-intervention
  Copenhagen Psychosocial Questionnaire (COPSOQ-II) long form; a battery of scales used in research to measure psychosocial factors at work (128-items total); 3-items using a 4-point Likert scale from 0, no not at all to 100, yes certainly
Psychosocial factors at work: trust regarding management | Baseline, pre-intervention
  Copenhagen Psychosocial Questionnaire (COPSOQ-II) long form; a battery of scales used in research to measure psychosocial factors at work (128-items total); 4-items using a 5-point Likert scale from 0, to a very small extent to 100, to a very large extent
Psychosocial factors at work: mutual trust between employees | Baseline, pre-intervention
  Copenhagen Psychosocial Questionnaire (COPSOQ-II) long form; a battery of scales used in research to measure psychosocial factors at work (128-items total); 3-items using a 5-point Likert scale from 0, to a very small extent to 100, to a very large extent
Psychosocial factors at work: justice and respect | Baseline, pre-intervention
  Copenhagen Psychosocial Questionnaire (COPSOQ-II) long form; a battery of scales used in research to measure psychosocial factors at work (128-items total); 4-items using a 5-point Likert scale from 0, to a very small extent to 100, to a very large extent
Psychosocial factors at work: social responsibility | Baseline, pre-intervention
  Copenhagen Psychosocial Questionnaire (COPSOQ-II) long form; a battery of scales used in research to measure psychosocial factors at work (128-items total); 4-items using a 5-point Likert scale from 0, to a very small extent to 100, to a very large extent
Psychosocial factors at work: self rated health | Baseline, pre-intervention
  Copenhagen Psychosocial Questionnaire (COPSOQ-II) long form; a battery of scales used in research to measure psychosocial factors at work (128-items total); 1-item using a 5-point Likert scale from 0, poor to 100, excellent
Psychosocial factors at work: burnout | Baseline, pre-intervention
  Copenhagen Psychosocial Questionnaire (COPSOQ-II) long form; a battery of scales used in research to measure psychosocial factors at work (128-items total); 4-items using a 5-point Likert scale from 0, not at all to 100, all the time
Psychosocial factors at work: stress | Baseline, pre-intervention
  Copenhagen Psychosocial Questionnaire (COPSOQ-II) long form; a battery of scales used in research to measure psychosocial factors at work (128-items total); 4-items using a 5-point Likert scale from 0, not at all to 100, all the time
Psychosocial factors at work: sleeping troubles | Baseline, pre-intervention
  Copenhagen Psychosocial Questionnaire (COPSOQ-II) long form; a battery of scales used in research to measure psychosocial factors at work (128-items total); 4-items using a 5-point Likert scale from 0, not at all to 100, all the time
Psychosocial factors at work: depressive symptoms | Baseline, pre-intervention
  Copenhagen Psychosocial Questionnaire (COPSOQ-II) long form; a battery of scales used in research to measure psychosocial factors at work (128-items total); 4-items using a 5-point Likert scale from 0, not at all to 100, all the time
Psychosocial factors at work: somatic stress symptoms | Baseline, pre-intervention
  Copenhagen Psychosocial Questionnaire (COPSOQ-II) long form; a battery of scales used in research to measure psychosocial factors at work (128-items total); 4-items using a 5-point Likert scale from 0, not at all to 100, all the time
Psychosocial factors at work: cognitive stress symptoms | Baseline, pre-intervention
  Copenhagen Psychosocial Questionnaire (COPSOQ-II) long form; a battery of scales used in research to measure psychosocial factors at work (128-items total); 4-items using a 5-point Likert scale from 0, not at all to 100, all the time
Psychosocial factors at work: perceived self-efficacy for life solving problems | Baseline, pre-intervention
  Copenhagen Psychosocial Questionnaire (COPSOQ-II) long form; a battery of scales used in research to measure psychosocial factors at work (128-items total); 6-items using a 4-point Likert scale from 0, does not fit to 100, fits perfectly
Psychosocial factors at work: conflicts and offensive behaviors | Baseline, pre-intervention
  Copenhagen Psychosocial Questionnaire (COPSOQ-II) long form; a battery of scales used in research to measure psychosocial factors at work (128-items total); 7-items using 5-point Likert scale from 0, no to 100, yes, daily
Occupational Self-efficacy for performing job-related duties | Baseline, pre-intervention
  Occupational Self-Efficacy Scale; 20-items rated using a 6-point Likert scale from 1, strongly disagree to 6, strongly agree
Organizational culture | Baseline, pre-intervention
  Competing Values Culture Assessment; 6-dimensions, 48-items assessing the present and future where the sum of 4-items per column (present; future) must equal 100; provides insight on how provider perceives the organization to be and must change to be in order to accomplish its highest objectives and goals

CONTACTS AND LOCATIONS:
Overall Officials: Abigail Gamble, PhD, MS, Principal Investigator — University of Mississippi Medical Center
Locations (1):
- Mississippi State Department of Health, Jackson, Mississippi, United States

IPD SHARING:
Plan to Share IPD: No
Given this is a single arm feasibility study with 20 participants, individual participant data will not be shared with other researchers.

REFERENCES:
- [Background] Gamble A, Baskin ML, Cranston KL, Herring SJ, Hinton E, Saulters MM, Moore JB, Welsch MA, Beech BM. Effects of eHealth interventions on physical activity and weight among pregnant and postpartum women and the sociodemographic characteristics of study populations: a systematic review protocol. JBI Evid Synth. 2020 Nov;18(11):2396-2403. doi: 10.11124/JBISRIR-D-19-00378. PMID 32813415
- [Result] Gamble A, Saulters MM, Cranston KL, Jones DW, Herring SJ, Beech BM. Recruitment, Retention, and Engagement Strategies for Exercise Interventions With Rural Antenatal Adolescents: Qualitative Interviews With WIC Providers. J Public Health Manag Pract. 2020 Sep/Oct;26(5):497-502. doi: 10.1097/PHH.0000000000001027. PMID 32732725
- [Result] Gamble A, Beech BM, Blackshear C, Cranston KL, Herring SJ, Moore JB, Welsch MA. Recruitment planning for clinical trials with a vulnerable perinatal adolescent population using the Clinical Trials Transformative Initiative framework and principles of partner and community engagement. Contemp Clin Trials. 2021 May;104:106363. doi: 10.1016/j.cct.2021.106363. Epub 2021 Mar 15. PMID 33737198
- [Result] Gamble A, Beech BM, Blackshear C, Herring SJ, Welsch MA, Moore JB. Changes in Physical Activity and Television Viewing From Pre-pregnancy Through Postpartum Among a Socioeconomically Disadvantaged Perinatal Adolescent Population. J Pediatr Adolesc Gynecol. 2021 Dec;34(6):832-838. doi: 10.1016/j.jpag.2021.06.009. Epub 2021 Jul 13. PMID 34271198